CLINICAL TRIAL: NCT01384084
Title: URINARY INCONTINENCE AND URO-GENITAL PROLAPSE: A RANDOMIZED TRIAL OF PELVIC ORGAN PROLAPSE REPAIR PLUS MINI-SLING VERSUS PELVIC ORGAN PROLAPSE REPAIR ALONE
Brief Title: Pelvic Organ Prolapse Repair Plus Mini-Sling Versus Pelvic Organ Prolapse Repair Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Luigi Mearini, senior assistant, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPerugia-1
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence
Keywords: pelvic organ prolapse; urinary incontinence; sacropexy; sling
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- POP repair plus mini-sling (Experimental): Patients affected by urogenital prolapse and urinary incontinence, who are candidates for pelvic organ prolapsed repair using sacropexy, will receive sacropexy plus anti-incontinence procedure (mini-sling).
  Interventions: Procedure: POP repair plus mini-sling
- pelvic organ prolapse repair (Active Comparator): Patients affected by urogenital prolapsed and urinary incontinence, who are candidates for pelvic organ prolapsed repair using sacropexy, will receive sacropexy alone.
  Interventions: Procedure: POP repair

INTERVENTIONS:
Procedure: POP repair plus mini-sling — For POP, the anterior vaginal wall is dissected from the bladder to expose a vaginal wall area where the mesh will be attached. The procedure is repeated for the posterior vaginal wall. The sacral promontory surface is prepared and 1 non-reabsorbable sutures are placed into the sacral periosteum.
  A mini sling system will be used, placing a urethral low-tension tape anchored to the obturator muscles bilaterally at the level of tendinous arc. This mini-sling is a polypropylene monofilament mesh.
  Arms: POP repair plus mini-sling
Procedure: POP repair — For POP repair, the anterior vaginal wall is dissected from the bladder to expose a vaginal wall area where the mesh will be attached. The procedure is repeated for the posterior vaginal wall. The sacral promontory surface is prepared and 1 non-reabsorbable sutures are placed into the sacral periosteum. The peritoneum is closed over the meshes.
  Arms: pelvic organ prolapse repair

SUMMARY:
The investigators have performed colposacropexy in women with uterovaginal prolapse for many years with satisfactory results.

This study was designed to compare whether, in the treatment of patients with uro-genital prolapse and urinary incontinence, the addition of a contemporary anti-incontinence procedure such as mini-sling is associated with a reduction of post-operative urinary incontinence (correction of pre-existent urinary incontinence and prevention of masked urinary incontinence).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by III-IV grade urogenital urogenital prolapsed and urinary incontinence
* Candidates for pelvic organ prolapsed repair using sacropexy
* Prospectively randomized, using a predetermined computer-generated randomization code (4 blocks), to sacropexy plus anti-incontinence procedure (mini-sling) or sacropexy alone

Exclusion Criteria:

* fertile patients
* contraindication to major surgery
* uterine cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
urinary incontinence | 12 months
  long-term relief of symptoms with anatomic correction of prolapse and subjective/objective correction of urinary incontinence

SECONDARY OUTCOMES:
peri and post-operative complications | 1 month
  Operative time and morbidity according to Clavien-Dindo classification, post-operative complications, length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Dept. University of Perugia, Perugia, Italy

REFERENCES:
- [Background] Costantini E, Lazzeri M, Bini V, Del Zingaro M, Zucchi A, Porena M. Pelvic organ prolapse repair with and without prophylactic concomitant Burch colposuspension in continent women: a randomized, controlled trial with 8-year followup. J Urol. 2011 Jun;185(6):2236-40. doi: 10.1016/j.juro.2011.01.078. Epub 2011 Apr 16. PMID 21497843
- [Background] Costantini E, Lazzeri M, Zucchi A, Bini V, Mearini L, Porena M. Five-year outcome of uterus sparing surgery for pelvic organ prolapse repair: a single-center experience. Int Urogynecol J. 2011 Mar;22(3):287-92. doi: 10.1007/s00192-010-1342-7. Epub 2010 Dec 9. PMID 21152903
- [Background] Novara G, Artibani W, Barber MD, Chapple CR, Costantini E, Ficarra V, Hilton P, Nilsson CG, Waltregny D. Updated systematic review and meta-analysis of the comparative data on colposuspensions, pubovaginal slings, and midurethral tapes in the surgical treatment of female stress urinary incontinence. Eur Urol. 2010 Aug;58(2):218-38. doi: 10.1016/j.eururo.2010.04.022. Epub 2010 Apr 23. PMID 20434257
- [Background] Costantini E, Lazzeri M, Bini V, Del Zingaro M, Zucchi A, Porena M. Burch colposuspension does not provide any additional benefit to pelvic organ prolapse repair in patients with urinary incontinence: a randomized surgical trial. J Urol. 2008 Sep;180(3):1007-12. doi: 10.1016/j.juro.2008.05.023. Epub 2008 Jul 17. PMID 18639302
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839